CLINICAL TRIAL: NCT04534283
Title: A Phase 2 Basket Trial of an ERK1/2 Inhibitor (LY3214996) in Combination With Abemaciclib for Patients Whose Tumors Harbor Pathogenic Alterations in BRAF, RAF1, MEK1/2, ERK1/2, and NF1.
Brief Title: A Basket Trial of an ERK1/2 Inhibitor (LY3214996) in Combination With Abemaciclib.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy.
Sponsor: Anita Turk (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Anita Turk, Assistant Professor of Clinical Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCC-0730
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cancer; Cancer Metastatic; BRAF V600E; MEK1 Gene Mutation; MEK2 Gene Mutation; ERK Mutation; RAF1 Gene Mutation
Keywords: Point Mutation; Metastatic Cancer; Advanced Cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — abemaciclib; LY3214996

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib + LY3214996 (Experimental): Subjects will receive Abemaciclib 150 mg orally twice daily with LY3214996 200 mg orally daily until disease progression, unacceptable toxicity, or patient preference to withdraw from study.
  Interventions: Drug: Abemaciclib; Drug: LY3214996

INTERVENTIONS:
Drug: Abemaciclib — Subjects will receive Abemaciclib 150 mg orally twice daily until disease progression, unacceptable toxicity, or patient preference to withdraw from study.
  Other Names: LY2835219
Drug: LY3214996 — Subjects will recieve LY3214996 200 mg orally daily until disease progression, unacceptable toxicity, or patient preference to withdraw from study.

SUMMARY:
The purpose of CTO-IUSCC-0730 study is to assess the clinical efficacy of LY3214996 in combination with abemaciclib at the recommended phase 2 dose of LY3214996 200 mg orally daily and abemaciclib 150 mg orally twice daily. Patients will be treated until evidence of disease progression, non-compliance with study protocol, unacceptable major toxicity, at subject's own request for withdrawal, or if the study closes for any reason.

ELIGIBILITY:
Inclusion Criteria:

Have a histological or cytological diagnosis of advanced unresectable or metastatic cancer (American Joint Committee on Cancer Staging Criteria) (Edge et al. 2009).

2. The patient must be, in the judgement of the investigator, an appropriate candidate for experimental therapy, either after available standard therapies (per available local guidelines) have failed to provide clinical benefit for their disease or after the patient has refused standard treatments.

3. Have one of the following alterations as defined below using a CLIA-certified next-generation sequencing test:

a. Point mutation in BRAF, RAF1, MEK1/2, or ERK1/2 that have been previously characterized to be gain-of-function mutations. These mutations have to be specified as gain-of-function as listed in the OncoKB and/or JAX-CKB databases. i. Patients with NSCLC that harbor BRAF V600E treated with prior RAF and/or MEK inhibition therapy will be excluded.

ii. Patients with tumor types other than NSCLC that harbor BRAF V600E mutations who have been treated and progressed on prior BRAF and/or MEK inhibition will be included.

iii. Patients with NSCLC that harbor BRAF V600E will only be enrolled if they are not a candidate for FDA approved therapy

1. Amplification of RAF1 defined as >6 copies of the respective gene.
2. Gene fusion in which BRAF, RAF1, MEK1/2, or ERK1/2, is a fusion partner; in which the fusion is determined to be in-frame; and the kinase domain of BRAF, RAF1, MEK1/2, or ERK1/2 is retained.
3. Point mutations, frameshift insertions/deletions, splice site mutations, or stop gain mutations that results in loss-of-function of NF1.

   4. Have measurable disease amenable to biopsy. If biopsy is deemed unsafe at time of procedure, patients will remain eligible for study.

   5. Must be able to provide written informed consent and HIPAA authorization for release of personal health information.

   6. Have a performance status (PS) of 0 or 1 on the Eastern Cooperative Oncology (Group (ECOG) scale (Oken et al. 1982) within 21 (+/-7) days prior to registration for protocol therapy.

   7. Have discontinued previous systemic treatments > 3 weeks for cancer prior to first dose of investigational therapy. Patient must have resolution, except for alopecia, of all clinically significant toxic effects of prior chemotherapy, surgery, or radiotherapy to Grade ≤1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.

   8. Have adequate organ function, as defined below: Laboratory Value (Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; ANC = absolute neutrophil count; ULN = upper limit of normal.) Hematologic ANC ≥1.5 × 109/L Platelets ≥100 × 109/L Hemoglobin ≥9.0 g/dL Transfusions to increase the patient's hemoglobin level to 9 g/dL are not permitted within 1 week prior to the baseline hematology profile Hepatic Total bilirubin ≤1.5 × ULN OR <2.0 mg/dL in patients with Gilbert's disease ALT and AST ≤2.5 × ULN OR ≤5 × ULN if the liver has tumor involvement Renal Serum creatinine OR Calculated creatinine clearance (see Appendix 3) ≤1.5 × ULN OR ≥50 mL/min

   9. Are at least 18 years old at the time of screening.

   10. Are male patients who are sterile (including vasectomy confirmed by post vasectomy semen analysis), or agree to use an effective method of contraception and not to donate sperm, or who practice total abstinence from heterosexual activity, starting with the first dose of study treatment, during the study, and for at least 6 months following the last dose of study treatment.

   11. Are female patients of non-childbearing potential (surgically sterile after having a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy or postmenopausal), or are female patients of child-bearing potential who are not pregnant, as confirmed by a serum pregnancy test within 14 (+/-7) days prior to receiving first dose of study treatment and who agree to use 2 methods of birth control (hormonal or intrauterine plus a barrier method) or practice total abstinence from heterosexual activity during the study for at least 6 months following the last dose of the study treatment.

   12. Are able to swallow capsules or tablets 13. Have an estimated life expectancy of ≥12 weeks, in the judgment of the investigator.

Exclusion Criteria:

1. Have a serious concomitant systemic disorder (for example, active infection or a gastrointestinal disorder causing clinically significant symptoms such as nausea, vomiting or diarrhea, or profound immune suppression) that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol.
2. Have or known activated/reactivated hepatitis A, B, or C (screening is not required).
3. Uncontrolled human immunodeficiency virus (HIV) infection are considered ineligible. HIV- infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

   Known HIV positive patients who meet the following criteria will be considered eligible:
   1. CD4 count ≥ 350 cells/mm3
   2. Undetectable viral load
   3. Maintained on modern therapeutic regimens utilizing non-CYP interactive agents (i.e. excluding ritonavir)
   4. No history of AIDS-defining opportunistic infections
4. Have symptomatic and untreated central nervous system (CNS) malignancy or metastasis (screening is not required).

   a. Patients with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids for their CNS metastasis and/or anticonvulsants. Patient must be > 4 weeks from therapy completion (including radiation and/or surgery) and clinically stable at time of study entry. Brain MRI or head CT is required at screening for patients with known brain metastases.
5. Have current hematologic malignancies, acute or chronic leukemia
6. Have a second primary malignancy that in the judgment of the principle investigator may affect the interpretation of results
7. Have prior malignancies within the last 3 years prior to study enrollment. Patients with carcinoma in situ of any origin and patients with prior malignancies who completed curative intent-treatment and whose likelihood of recurrence is very low, as judged by the principal investigator, will remain eligible for this study. The principal investigator will approve enrollment of patients with prior malignancies in remission before these patients are enrolled.
8. Are currently enrolled in a clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
9. Have participated, within the last 28 days in a clinical trial involving an investigational product.
10. Have previously completed or withdrawn from this study or any other study investigating an ERK1/2 inhibitor.
11. Had prior therapy with an ERK1/2 inhibitor.
12. Had prior chemotherapy within 3 weeks of study registration.
13. Had prior non-CNS radiation within 2 weeks of study registration. Please refer to exclusion criteria #4 for patients who have required radiation for CNS disease.
14. If female, is pregnant, breastfeeding, or planning to become pregnant.
15. Currently using concomitant medications that are strong inhibitors or inducers of CYP3A4.
16. Have serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.

    1. This includes cardiogenic syncope, ventricular arrhythmias, history of sudden cardiac arrest, or severe dyspnea at rest or requiring oxygen therapy.
    2. This includes patients with any evidence of interstitial lung disease (ILD) (not just serious and/or uncontrolled ILD) and any history of severe ILD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Turk, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital / IU Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abemaciclib + LY3214996
Started | 16
Completed | 0
Not Completed | 16
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Disease Progression | 12
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients who received at least one dose of study treatment.
Arm/Group | Abemaciclib + LY3214996
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Performance Status (ECOG) at screening [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) measures how the disease impacts a patient's daily living abilities. Lower scores are considered better.
  0=Fully active, able to carry on all pre-disease performance without restriction
  1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 3
    1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The number of patients who achieve a best overall response of complete response (CR) or partial response (PR) divided by the total number of patients treated (efficacy population) as determined by RECIST v1.1.
Time Frame: from cycle 1 day 1 until safety follow up visit (up to 1 year)
Population: All enrolled patients who received at least one dose of study treatment and had a post-baseline imagining.
Measure: Number; unit: percentage of patients
Arm/Group | Abemaciclib + LY3214996
Number analyzed (Participants) | 12
percentage of patients | 0

2. Secondary Outcome: Number of Patients With Treatment Related Adverse Events Grade 3 or Above
Description: Number of unique patients with any Abemaciclib or LY3214996 treatment related (possible, probable, or definite) adverse events with grade >=3. CTCAE Version 5.0 will be used.
Time Frame: baseline until safety follow up visit (up to 1 year)
Population: All enrolled patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib + LY3214996
Number analyzed (Participants) | 13
Participants | 6

3. Secondary Outcome: Duration of Overall Response Rate
Description: Measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented through RECIST v1.1. Please note that there were no patients who achieved Complete Response (CR) or Partial Response (PR) within this study.
Time Frame: up to 1 year
Population: All enrolled patients who received at least one dose of study treatment and had post-baseline imaging.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Abemaciclib + LY3214996
Number analyzed (Participants) | 12
days | 0 [0 to 0]

4. Secondary Outcome: Progression Free Survival
Description: The time from the date of start of treatment to the first date of the observed clinical or radiologically documented PD or death due to any cause, whichever occurs first. For patients who are not known to have died or progressed as of the data-inclusion cut-off date, PFS time will be censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systematic anticancer therapy. Assessment are completed using RECIST v1.1. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated.
Time Frame: up to 1 year, 1 month
Population: All enrolled patients who received at least one dose of study treatment and had a post-baseline imagining.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib + LY3214996
Number analyzed (Participants) | 12
months | 2.1 [1.6 to 7.6]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: All enrolled patients who received at least one dose of study treatment were included in the Adverse Events summaries (this includes the Serious Adverse Events). Patients who did not receive any study drug were not included.
Arm/Group | Abemaciclib + LY3214996
All-Cause Mortality (participants affected / at risk) | 10/13
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib + LY3214996 (N=13)
Anemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib + LY3214996 (N=13)
Anemia (Blood and lymphatic system disorders) | 5
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Anal hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Rectal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 1
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 10
Fever (General disorders) | 4
Pain (General disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to smaller number of patients enrolled than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT04534283/Prot_SAP_000.pdf